CLINICAL TRIAL: NCT00004112
Title: A Phase III Randomized Trial of CHOP Chemotherapy Plus Rituxan (IDEC-C2B8) Versus CHOP Chemotherapy Alone for Newly Diagnosed, Previously Untreated, Aggressive Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy With or Without Rituximab in Treating Patients With Newly Diagnosed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 0447-97-FB; P30CA036727 (NIH); UCLA-HSPC-9812071 (Other: University of California - Los Angeles); NCI-G99-1601 (Other Grant/Funding Number: National Cancer Institute (NCI))
Record Dates: First submitted 1999-12-10; First posted 2004-05-25 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Lymphoma
Keywords: stage II adult diffuse small cleaved cell lymphoma; stage II adult diffuse mixed cell lymphoma; stage II adult diffuse large cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; anaplastic large cell lymphoma; stage II mantle cell lymphoma; stage II small lymphocytic lymphoma; stage II marginal zone lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; VAP-cyclo protocol; Cyclophosphamide; Vincristine; Doxorubicin; Prednisolone; Drug Therapy; liposomal doxorubicin; Prednisone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: rituximab
  Other Names: Rituxan
Drug: CHOP regimen — Cyclophosphamide, vincristine and doxorubicin as a drip into the bloodstream (intravenously) and prednisolone (steroid) as tablets taken with or after food.
  Other Names: cyclophosphamide, vincristine, doxorubicin, prednisolone
Drug: cyclophosphamide
  Other Names: chemotherapy
Drug: doxorubicin hydrochloride
  Other Names: Lipodox, Lipodox 50, and Doxil
Drug: prednisone
  Other Names: Prednisone Intensol, Deltasone, Rayos, steroid
Drug: vincristine sulfate
  Other Names: Oncovin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known whether combination chemotherapy plus rituximab is more effective than combination chemotherapy alone for non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without rituximab in treating patients who have newly diagnosed non-Hodgkin's lymphoma that has not been treated previously.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether the addition of rituximab to cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) increases the failure-free survival of patients with newly diagnosed, previously untreated, aggressive B-cell non-Hodgkin's lymphoma. II. Determine whether the addition of rituximab changes the toxicity profile attributed to CHOP chemotherapy in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center, histology (diffuse small cleaved cell, diffuse mixed, and diffuse large cell vs immunoblastic large cell, mantle cell, and marginal zone), and risk group (low vs intermediate vs high). Patients enter one of two treatment arms: Arm I: Patients receive rituximab IV on day 1, followed by cyclophosphamide IV, doxorubicin IV, vincristine IV, and oral prednisone for 5 consecutive days beginning on day 3. Arm II: Patients receive cyclophosphamide IV, doxorubicin IV, vincristine IV, and oral prednisone daily for 5 consecutive days beginning on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients will be followed for 3 years.

PROJECTED ACCRUAL: A total of 270 patients (135 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed, aggressive (stage II-IV) B-cell non-Hodgkin's lymphoma, including but not limited to:

  * Mantle cell
  * Diffuse large cell
  * Diffuse mixed cell
  * Anaplastic large cell (B-cell type)
  * Diffuse small cleaved cell
  * Marginal zone lymphoma
  * CD20 positive
* 19 years old and over
* WHO 0-2
* Karnofsky 70-100%
* Life expectancy at least 6 months
* Absolute neutrophil count greater than 1,000/mm3 (unless due to non-Hodgkin's lymphoma (NHL) bone marrow involvement)
* Bilirubin less than 3.0 mg/dL
* Alkaline phosphatase less than 3 times upper limit of normal (ULN)
* SGOT less than 3 times ULN
* Fertile patients must use effective contraception
* HIV negative
* Nonsteroidal hormones for non-lymphoma related conditions allowed (e.g., insulin for diabetes)

Exclusion Criteria:

* No prior T-cell lymphoma
* Not pregnant or nursing
* No other serious disease or medical condition that would interfere with compliance
* No other concurrent chemotherapy
* No concurrent corticosteroids (unless for prevention of nausea or vomiting)
* No concurrent radiotherapy No other concurrent investigational agents

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09-01 (Actual); Primary Completion 2000-12-01 (Actual); Study Completion 2003-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Study Chair — University of Nebraska
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - University of Nebraska Medical Center, Omaha, Nebraska